CLINICAL TRIAL: NCT00882934
Title: A Single-Blind, Controlled, Randomized, Parallel-Group Study of the Efficacy of Patients' Awareness on the Composition of the Experimental Drug in the Treatment of Erectile Dysfunction.
Brief Title: The Management of Erectile Dysfunction With Placebo Only
Acronym: DAFA06
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Eloisio Alexsandro da Silva, Service of Urology. Laboratory for Translational Research in Urology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DAFA06
Record Dates: First submitted 2009-04-15; First posted 2009-04-17 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Impotence; Erectile Dysfunction
Keywords: Placebo; Placebo Effect; Sexual Dysfunction; Erectile Dysfunction; Clinical Trial
MeSH Terms: conditions — Erectile Dysfunction; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A1 (Experimental): Arm 1 received an informative letter explaining that they were allocated to receive a substance for Erectile Dysfunction treatment.
  Interventions: Other: Induction to efficient treatment
- A2 (Placebo Comparator): Arm 2 (A2) was written informed that they could or could not receive an active drug for ED treatment.
  Interventions: Other: Doubt to the efficacy of treatment
- A3 (Experimental): Arm 3 (A3) was properly written informed to be using no effective drug for ED treatment.
  Interventions: Other: Induction to ineffective treatment

INTERVENTIONS:
Other: Induction to efficient treatment — Informative letters.
  Arms: A1
Other: Doubt to the efficacy of treatment — Informative letters.
  Arms: A2
Other: Induction to ineffective treatment — Informative letters
  Arms: A3

SUMMARY:
Placebo-controlled randomized clinical trials (RCT) are the gold standard to provide applicable evidence for clinical practice. A vast number of RCTs for treatment of several disorders has shown a mean placebo effect of 30%. Erectile dysfunction (ED) is a high prevalent disease and its first-line therapy is oral phosphodiesterase type-5 inhibitor (iPDE5) (i.e., sildenafil, vardenafil and tadalafil). Although the placebo effect in iPDE5 RCT occurred at a rate as high as 50%, in the last decade, with the revolutionary discovery of effective pharmacotherapy for ED, oral iPDE5 has become one of the most common prescribed drugs for men. The objective of this study is to evaluate the influence of patients' awareness on the composition of the therapeutic drug in the outcomes of the oral treatment for ED.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Complaint of ED for at least 6 months prior the start of the study, according to medical history and to the questionnaires IIEF, SEAR and QEQ.
* A stable heterosexual relationship.
* To be in good health prior the participation in the study, with no important clinical abnormalities, determined by: clinical history, physical examination, blood chemistry and hematology, urinalysis (If the standard values of the laboratory for these tests are not evidenced, subjects can be included if the researcher consider the changes as not clinically significant).

Exclusion Criteria:

* History of significant cardiovascular, pulmonary, gastrointestinal, hematological, neurological (including epilepsy), locomotor, immunologic, ophthalmic, metabolic, endocrine, thromboembolic, rheumatologic, cancer, kidney or liver disease.
* Diagnosis of psychiatric conditions, e.g. depression, anxiety, dysthymia, mania, panic, agoraphobia, social phobia, suicidal ideation, obsessive-compulsive disorder, post-traumatic stress, psychotic disorders, schizophrenia, alcoholism, dependence on psycho-active substances.
* History of HIV, hepatitis B or hepatitis C.
* Hyperprolactinemia or untreated hypothyroidism.
* Any condition, which, in the opinion of the investigator, may interfere with the participation of the subject in the study (e.g. difficulty to meet the requirements of the study, attend the consultations, answer the questionnaires).
* Report of significant clinical problems by the subject's partner, such as decreased sexual interest, pain during relations or other forms of sexual dysfunction that interfere in the relationship with the sexual partner.
* Patient or partner willing to undergo a surgical procedure during the study period, which may interfere in the results.
* Peyronie's disease, which may lead to impossibility to penetrate or cause pain during the sexual intercourse.
* Use of nitrates.
* Illiterate patient.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2006-10; Primary Completion 2007-10 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
IIEF erectile function domain score | 4 AND 8 Weeks
Quality of Erection Questionnaire (QEQ) | 4 and 8 weeks

SECONDARY OUTCOMES:
IIEF orgasmic function, sexual desire, intercourse satisfaction and overall satisfaction domain scores | 4 and 8 weeks
SEAR questionnaire | 4 and 8 weeks
EDITS questionnaire | 4 and 8 weeks
GEAQ questionnaire | 4 and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eloisio Alexsandro da Silva, MD, PhD, Study Chair — Laboratory for Translational Research in Urology